CLINICAL TRIAL: NCT04755166
Title: Lateral Ridge Augmentation With Two Different Compositions of Deproteinized Bovine Bone and Autogenous Bone: A Randomized, Controlled Study
Brief Title: Horizontal Augmentation With Deproteinized Bovine Bone Mineral Alone or in Combination With Particulate Autogenous Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NU-Hospital Organization, Sweden (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Hanna Aludden, Principal Investigator, NU-Hospital Organization, Sweden
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LRA humans
Record Dates: First submitted 2021-02-07; First posted 2021-02-15 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Edentulous Jaw
Keywords: Bone substitutes; Imaging-Three-Dimensional; alveolar ridge augmentation; dental implants; Bio-Oss; Guided bone regeneration
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- 100:0 (Experimental): 100 % bone substitute, 0% autogenous bone
  Interventions: Procedure: Lateral ridge augmentation
- 90:10 (Experimental): 90% bone substitute, 10% autogenous bone
  Interventions: Procedure: Lateral ridge augmentation

INTERVENTIONS:
Procedure: Lateral ridge augmentation

SUMMARY:
Background: Placement of oral implants is frequently compromised due to atrophy of the alveolar process. Lateral ridge augmentation with an autogenous bone block is frequently necessary to increase the width of the alveolar process before implant installation. However, harvesting of an autogenous bone block is associated with donor site morbidity. Consequently, bone substitutes alone or in combination with particulate autogenous bone graft are used increasingly to simplify the surgical procedure. Animal and human studies evaluating lateral ridge augmentation with Bio-Oss alone or in combination with particulate autogenous bone graft have demonstrated new bone formation and high implant survival. However, the optimal ratio of Bio-Oss and particulate autogenous bone graft for lateral ridge augmentation and long-term implant survival is unknown.

Purpose: Test the H0-hypothesis of no difference in long-term implant survival, newly formed bone, volumetric stability of the graft, gained width of the alveolar process and patient satisfaction after lateral ridge augmentation with Bio-Oss alone or in combination with a diminutive amount of autogenous bone graft.

Material and methods: lateral ridge augmentation will be performed in 20 adults with two different ratios of Bio-Oss and autogenous bone graft after a split mouth design. Clinical and radiological measurements will evaluate the long-term implant survival. Cone beam computer tomography (CBCT) will be obtained preoperatively, immediately postoperatively, prior to implant placement, 2 years after implant installation and 5 years after implant installation to estimate the volumetric changes of the augmented area. Moreover, the amount of newly formed bone will be estimated by histologic evaluation after implant placement.

Conclusion: Long-term implant survival has never been evaluated after lateral ridge augmentation with Bio-Oss alone or in combination with a diminutive amount of autogenous bone graft.

ELIGIBILITY:
Inclusion Criteria:

* Total or partial bilateral edentulism
* Horizontal bone width less than 4 mm at planned sites of implant installation or need of augmentation of aesthetic reasons for optimal implant placement

Exclusion Criteria:

* Uncontrolled systematic disease
* History of radiation in the area
* Smoking habits (free of smoking habits more than 1 month prior to treatment)
* Treatment with bisphosphonates
* Patients who cannot complete the 5-year observation period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Newly formed bone | 10 months after treatment
  Amount of newly formed bone in the graft assessed by histological measurements
Height in mm | 10 months after treatment
  Height of the augmented area assessed by radiological measurements
Volume in mm3 | 10 months after treatment
  Volume of the augmented area assessed by clinical and radiological measurements
Implant survival | 1 year after placement of the implants
  Survival of implants placed in the graft assessed by clinical and radiological measurements
Implant survival | 3 year after placement of the implants
  Survival of implants placed in the graft assessed by clinical and radiological measurements
Implant survival | 5 year after placement of the implants
  Survival of implants placed in the graft assessed by clinical and radiological measurements

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Aludden, DDS, PhD, Principal Investigator — NU Hospital Organisation, Trollhättan, Sweden
Locations (1):
- NU Hospital Organization, Trollhättan, Sweden